CLINICAL TRIAL: NCT05735080
Title: A Phase 1/2, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of INX-315 in Patients With Advanced Cancer
Brief Title: Open-Label Study to Evaluate the Safety, Tolerability, PK, and Efficacy of INX-315 in Patients With Advanced Cancer
Acronym: INX-315-01
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Incyclix Bio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INX-315-01
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Breast Cancer Metastatic; Hormone Receptor Positive Tumor; Human Epidermal Growth Factor 2 Negative Carcinoma of Breast; Ovarian Cancer; CCNE1 Amplification; Solid Tumor; Advanced Cancer; Metastatic Cancer
Keywords: CDK2; CDK4/6i; cyclin dependent kinase 2; CCNE1
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Neoplasm Metastasis | interventions — Fulvestrant; abemaciclib

STUDY DESIGN:
Intervention Model Description: Part A will be a dose escalation guided by BOIN design for treatment assignment and dosing rules.
  Part B will be dose expansion, patients will be randomly assigned to receive one of the identified doses of INX-315 in monotherapy
  Part C will be dose expansion, patients will receive INX-315 in combination treatment with abemaciclib and fulvestrant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: Dose Escalation (Experimental): Multiple doses of INX-315 monotherapy, oral administration
  Interventions: Drug: INX-315
- Part B: Ovarian Dose Expansion (Experimental): INX-315 monotherapy, oral administration
  Interventions: Drug: INX-315
- Part C: HR+/HER2- BC Dose Expansion (Experimental): INX-315 in combination with abemaciclib (oral administration) and fulvestrant (IM)
  Interventions: Drug: INX-315; Drug: Fulvestrant; Drug: Abemaciclib
- Part A INX-315 + Fulvestrant (Experimental): INX-315 dose plus Fulvestrant 500mg (IM)
  Interventions: Drug: INX-315; Drug: Fulvestrant

INTERVENTIONS:
Drug: INX-315 — Oral administration
Drug: Fulvestrant — Fulvestrant will be combined with INX-315
  Other Names: faslodex
  Arms: Part A INX-315 + Fulvestrant; Part C: HR+/HER2- BC Dose Expansion
Drug: Abemaciclib — Abemaciclib will be combined with INX-315
  Other Names: Verzenio
  Arms: Part C: HR+/HER2- BC Dose Expansion

SUMMARY:
Incyclix Bio (Incyclix) is developing INX-315 as an oral, small molecule inhibitor of cyclin dependent kinase 2 (CDK2) for the treatment of human cancers. This first-in-human study is designed to evaluate the safety, tolerability, pharmacokinetics (PK) and preliminary antitumor activity of INX-315 in patients with recurrent advanced/metastatic cancer, including hormone receptor positive (HR+)/Human Epidermal Growth Factor Receptor 2 Negative (HER2-) breast cancer who progressed on a prior cyclin-dependent kinase 4/6 inhibitor (CDK4/6i) regimen, and CCNE1-amplified solid tumors who progressed on standard of care treatment. The study will be conducted in 3 parts: Part A (INX-315 monotherapy dose escalation and combination therapy with fulvestrant), Part B (ovarian cancer INX-315 monotherapy dose expansion), and Part C (INX-315 combination therapy with abemaciclib [a CDK4/6i] and fulvestrant [a SERD] in advanced/metastatic breast cancer; dose escalation and expansion).

DETAILED DESCRIPTION:
Study INX-315-01 is a first-in-human, Phase 1/2, open-label, dose escalation and dose-expansion study to evaluate the safety, PK, and preliminary antitumor activity of INX-315 in patients with advanced/metastatic cancers. The study will be conducted in 3 parts: Part A (dose escalation and combination therapy) and Part B (ovarian cancer dose expansion) and Part C (breast cancer dose escalation lead-in and expansion).

Part A is the dose-escalation portion of the study to evaluate the safety, tolerability, and PK of INX-315 monotherapy. Dosing decisions will be guided using a Bayesian optimal interval (BOIN) design. Up to 60 patients with recurrent advanced/metastatic cancer, including patients with HR+/HER2- breast cancer who progressed on a prior CDK4/6i regimen, and solid tumors, including ovarian cancer with known amplification of CCNE1 are planned to be enrolled in Part A.

Dose-limiting toxicities (DLTs) will be assessed during the first treatment cycle, i.e., the first 28 days of treatment (the DLT period). Patients who are evaluable for DLT assessment are those patients who are enrolled, received >=80% of the planned study drug doses during the DLT assessment period, and complete the 28-day DLT period.

Additionally, Part A will have two cohorts that will include INX-315 plus fulvestrant in HR+/HER2- patients who have have had prior treatment with CDK4/6i.

Part B will expand at least two dose levels determined by the SMC. Part B will enroll patients with platinum-refractory or platinum-resistant advanced/ metastatic ovarian cancer patients with CCNE1 amplifications. Part B will open for enrollment once the SMC has selected the dose levels to be evaluated from the Part A portion of the study. Part A patients cannot re-join or continue the study in Part B. Approximately 30 patients will be equally randomized to receive one of the dose levels of INX-315.

Part C will be an expansion cohort, patients with HR+/HER2- breast cancer will be enrolled in this cohort. Patients will receive INX-315 along with abemaciclib and fulvestrant. Approximately 50 patients will be enrolled in Part C.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced unresectable or metastatic ER+/HER2- BC that has progressed following treatment with a CDK4/6 inhibitor
2. Advanced/ metastatic platinum-resistant or platinum-refractory epithelial ovarian cancer (including fallopian tube cancer/primary peritoneal cancer) CCNE-1 amplified tumors that progressed after standard systemic therapy
3. Advanced or metastatic solid tumor with known amplification of CCNE-1 that has progressed after standard therapy, been intolerant to or is ineligible for standard therapy
4. At least one measurable lesion as defined by RECIST v1.1 that has not previously been irradiated
5. ECOG performance status score of 0 or 1.
6. Adequate organ function as demonstrated by the following laboratory values:

   1. Hemoglobin ≥ 9.0 g/dL
   2. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L
   3. Platelet count ≥ 100 × 109/L
   4. Estimated glomerular filtration rate (eGFR) of ≥60 mL/min
   5. Part A and B: Total bilirubin ≤ 1.5 × ULN; AST and ALT ≤ 2.5 × ULN; ≤ 5 × ULN in the presence of liver metastases Part C: Patients with GIlbert's syndrome with a total bilirubin ≤ 2.0 × ULN and direct bilirubin within normal limits
7. Negative pregnancy test

Exclusion Criteria:

1. Have received previous therapy with a CDK2/4/6 inhibitor or CDK2 inhibitor.
2. Have central nervous system (CNS) metastases or spinal cord compression that is associated with progressive neurological symptoms or requires corticosteroids (within 4 weeks of enrollment) to control the CNS disease.
3. Have known intracranial hemorrhage and/or bleeding diatheses.
4. Have visceral crisis, lymphangitic spread, or leptomeningeal carcinomatosis.
5. Have clinically active ongoing interstitial lung disease (ILD) of any etiology, including drug-induced ILD, and radiation pneumonitis within 28 days prior to initiation of study treatment.
6. Resting QTcF > 470 msec, a history of prolonged QT syndrome or Torsades de pointes, or a familial history of prolonged QT syndrome.
7. Uncontrolled, cardiovascular disease (including hypertension) with or without medication
8. History of other malignancies, except for the following: (1) adequately treated basal or squamous cell carcinoma of the skin; (2) curatively treated a) in situ carcinoma of the uterine cervix, b) prostate cancer, or c) superficial bladder cancer; or (3) other curatively treated solid tumor with no evidence of disease for ≥ 3 years.
9. Known HIV infection, including AIDS-related illness, or have active, uncontrolled infection (viral, bacterial, or fungal), including tuberculosis, hepatitis B virus, hepatitis C virus, or COVID-19 infection (symptoms and a positive test result).
10. Requires treatment with a prohibited medication or herbal remedy that cannot be discontinued at least 2 weeks before the start of study drug administration.
11. Have planned or anticipation of the need for major surgical procedure within 28 days of the first dose of study drug (procedures such as central venous catheter placement, tumor needle biopsy, and feeding tube placement are not considered major surgical procedures).
12. Unwilling or unable to comply with scheduled visits, study drug administration plan, laboratory tests, or other study procedures and study restrictions.
13. Radical radiotherapy within 28 days prior to study entry or palliative radiotherapy within 2 weeks prior to study entry.
14. Systemic anti-cancer therapy within 28 days or at least 5 half-lives, whichever is less, prior to the first dose of the study drug
15. Prior irradiation to > 25% of the bone marrow
16. Previous high-dose chemotherapy requiring prior stem cell transplant
17. Participation in other studies involving investigational drug(s) within 4 weeks prior to study entry.
18. Known or suspected hypersensitivity to active ingredient/excipients in INX-315 or fulvestrant or abemaciclib.
19. Known difficulty in swallowing or tolerating oral medications, or conditions which would impair absorption of oral medications such as active inflammatory gastrointestinal disease, uncontrolled nausea or vomiting (i.e., CTCAE ≥ Grade 3 despite antiemetic therapy), ongoing gastrointestinal obstruction/motility disorder/active inflammation, malabsorption syndrome, chronic diarrhea, known diverticular disease or previous gastric resection or lap band surgery.
20. Has a serious and/or uncontrolled pre-existing medical condition(s) that, in the judgment of the Investigator or the Sponsor, would preclude participation in this study (for example but not limited to, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Part A and B: Evaluate the incidents of treatment emergent adverse events and laboratory abnormalities in INX-315 monotherapy and in combination with fulvestrant | Up to 12 months
Part A: Evaluate the occurrence of dose-limiting toxicities (DLTs) during Cycle 1 | 28 days
Part A: Recommend at least two doses of INX-315 to be evaluated in the expansion phase | Up to 12 months
Part B: Overall response rate (ORR) | Up to 36 months
Part B: Selection of Recommended Phase 2 Dose (RP2D) | Up to 36 months
Part C Evaluate the incidents of treatment emergent adverse events and laboratory abnormalities for patients in combination treatment (INX_315+abemaciclib+fulvestrant) | Up to 12 months
Part C - Evaluate the antitumor activity of INX-315 in combination with abemaciclib and fulvestrant | Up to 12 months

SECONDARY OUTCOMES:
Characterize the maximum plasma concentration (Cmax) | Cycle 1 Day 1 and Day 15
Characterize the time to maximum plasma concentration (Tmax) | Cycle 1 Day 1 and Day 15
Characterize the Area under the plasma concentration versus time curve from time 0 to the end of the dosing interval (AUC0-24h) | Cycle 1 Day 1 and Day 15
Characterize the terminal half-life (t1/2) | Cycle 1 Day 1 and Day 15
Characterize the oral clearance (CL/F) | Cycle 1 Day 1 and Day 15
Part A: Overall response rate (ORR) | Up to 36 months
Disease control rate (DCR) | Up to 36 months
Progression free survival (PFS) | Up to 36 months
Duration of response (DOR) | Up to 36 months
Time to progression (TTP) | Up to 36 months
Overall survival (OS) | Up to 36 months
Part C Determine recommended dose of INX-315 in combination treatment for further study | Up to 12 months

CONTACTS AND LOCATIONS:
Locations (17):
- United States (15):
  - Florida Cancer Specialists, Lake Mary, Florida
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - Levine Cancer Institute (LCI)- Atrium Health, Charlotte, North Carolina
  - Duke Cancer Center/ DUMC, Durham, North Carolina
  - Gabrail Cancer Research Center, Canton, Ohio
  - Next Oncology, Dallas, Texas
  - UTSW Medical Center, Dallas, Texas
  - Oncology Consultants, Houston, Texas
  - Next Oncology, Houston, Texas
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
- Australia (2):
  - Peter MacCallum Cancer Center, Parkville, Victoria
  - Mater Hospital, South Brisbane

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: Data will be shared at the completion of the study, expected release date will be in 2026.